CLINICAL TRIAL: NCT03630861
Title: Establishment of a Signature of Circulating microRNA as a Tool to Aid Diagnosis of Primary Brain Tumors in Adults
Acronym: MIRNA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 14007; 2015-A00503-46 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-04-10; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-04

CONDITIONS: Brain Tumors
Keywords: MicroRNAs; Glioblastoma; nonglial tumors; stroke; diagnosis
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Stroke; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples aliquoted and stored may be used either for re-analysis if necessary for the current study or as part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- GBM: Primary glioblastoma (GBM)
- PCNSL: Primary CNS lymphomas (PCNSL)
- Brain metastases: Brain metastases (BM)
- Cerebral Stroke: Cerebral Stroke (CS)
- Healthy Volunteers: Healthy Volunteers (HV)

SUMMARY:
MIRNA is a prospective multi-center observational study designed to explore 762 plasma microRNAs in patients with malignant CNS tumours: 60 primary glioblastoma (GBM), 20 primary CNS lymphomas and 40 brain metastases in an attempt to establish plasma microRNA signatures specific to GBM capable of distinguishing them from malignant non-glial brain tumours. 20 patients with cerebral stroke and 20 healthy volunteers will also participate in the study, and for each patient, a panel of 762 microRNAs will be screened in plasma.

DETAILED DESCRIPTION:
Neuro-oncology faces two challenges: establishing an accurate, rapid diagnosis and having early therapeutic response. This applies particularly to glioblastoma (GBM) since the positive diagnosis is evoked on MRI imaging and the diagnosis of certainty provided by anatomopathology. There are no perfect techniques and there are problems of differential diagnosis in imaging. Sometimes the context does not allow biopsy or excision.

This study is a prospective multi-center observational study designed to be conducted in patients with malignant CNS tumours: primary glioblastoma (60 GBM), primary CNS lymphomas (20 PCNSL), brain metastases (40 BM), in an attempt to establish plasma microRNA signatures characteristic of a tumour process. Patients with cerebral stroke (20 CS) and healthy volunteers (20 HV) will also participate in the study. For each patient, a panel of 762 microRNAs will be screened in plasma.

First, the investigators will focus on the potentially diagnostic nature of the signature, which may prove useful when there are problems of differential diagnosis in imaging or when the context does not permit biopsy or excision. The main objective of the study is to establish a plasma microRNA signature specific to GBM, capable of distinguishing them from malignant non-glial brain tumours (PCNSL and BM). Within the main objective, discrimination will be established between GBM and malignant non-glial brain tumours.

Secondly, the quantitative approach of plasma miRNoma with 752 microRNAs studied in the different patient groups will allow for other objectives:1/ Establish plasma microRNA signatures characteristic of other types of brain tumours; 2/ Identify a plasma microRNA signature characteristic of the cerebral injury component independently of the tumor component with the CS and HV groups; 3/ Identify plasma microRNA signatures characteristic of GBM subtypes in relation to their genomic alterations; 4/ Establish correlations between plasma microRNA expression levels and data collected through multi-modality MRI imaging and anatomopathology.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria applicable to all study subject: adults aged between 50 and 75, affiliated to social protection and having signed a consent form.
2. Inclusion criteria for patients with a brain tumor (GBM, PCNSL): patients with clinical symptomatology and imaging suggestive of brain tumor, for whom a biopsy will be performed to make the diagnosis of certainty
3. Inclusion criteria for patients with BM: a priori asymptomatic patients who received treatment by stereotactic radiosurgery (gamma-knife) for small circumscribed BM (diameter < 3cm, less than 3)
4. Inclusion criteria for patients with CS: patients with clinical symptoms and imaging suggestive of acute stroke (< 24 hours, NIHSS score >5)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Brain tumors: GBM, PCNSL, BM
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
QR (relative amount) | Up to 3 months after the end of all samplings.
  QR (relative amount) of each plasma microRNA for GBM and non-glial tumors (PCNSL, BM).

SECONDARY OUTCOMES:
QR value of each microRNA for all groups | Up to 3 months after the end of all samplings
  QR value of each microRNA for all groups
Genetic abnormalities | Up to 3 months after the end of the study
  Genetic abnormalities of GBM subtypes
Main imaging and anatomopathology characteristics | Up to 3 months after the end of the study
  Description of main imaging and anatomopathological characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France